CLINICAL TRIAL: NCT04666519
Title: Are Zonulin Levels Associated With a Higher Risk of Infection?
Brief Title: Zonulin Biomarker for Diagnosis of Hip and Knee Infections
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: JPAR06D.229
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Surgical Site Infection; Zonulin
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Zonulin Biomarker — During revision hip and knee surgery, discarded fluid/blood will be tested for the presence of zonulin biomarkers

SUMMARY:
Prior studies investigating the etiopathogenesis of surgical site infection (SSI) traditionally suggested three main ways for the infection to occur: local contamination occurring during the surgery, hematogenous translocation of bacteria during concomitant bacteraemia, and contamination from adjacent infected tissues by the progression of the infective process. While most of the research on SSI focused on minimizing any source of pathogens at the time of the surgery, emerging evidence shows how acute and chronic SSI can emerge more often from bacteraemia or other tissues in the body, such as the gastrointestinal system, especially when dysbiosis and high permeability are retrieved.

Intercellular tight junctions (TJs) tightly regulate paracellular antigen trafficking. TJs are extremely dynamic structures that operate in several critical functions of the intestinal epithelium under both physiological and pathological circumstances. This paradigm was subverted in 1993 by the discovery of zonula occludens 1 (ZO-1) as the first component of the TJ complex 11 now being comprised of more than 150 proteins, including occludin, claudins, junctional adhesion molecules (JAMs), tricellulin , and angulins . However, despite major progress in our knowledge on the composition and function of the intercellular TJ, the mechanisms by which they are regulated are still incompletely understood. One of the breakthroughs in understanding the role of gut permeability in health and disease has been the discovery of zonulin, and the only physiologic intestinal permeability modulator described so far.

Since then, zonulin has been used as a marker for increased intestinal permeability and associated with soluble CD14 (sCD14) and lipopolysaccharide (LPS), other common markers associated with surgical complication, inflammation, and bacterial translocations.

As such, Zonulin could be a biomarker for mid- and long-term complications after total joint replacement such as infection, loosening, and mechanical complications associated with painful symptomatology.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent primary or aseptic revision total hip and knee arthroplasty.
* Patients who underwent revision total hip and knee arthroplasty for infective reasons
* Patients 18 years of age or older

Exclusion Criteria:

- Patients younger than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are undergoing a primary or aseptic revision total hip or knee replacement and patients who are having a revision hip or knee replacement for infection
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Infection Diagnosis | 90 days
  Zonulin levels will be tested on discarded blood/fluid during revision hip or knee replacement to see if there is a correlation between the zonulin levels and the development of an infection after their surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States